CLINICAL TRIAL: NCT03060720
Title: Systematic Hereditary Pancreatic Cancer Risk Assessment and Implications for Personalized Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew B. Yurgelun, MD, Matthew B. Yurgelun, MD, Dana-Farber Cancer Institute
Other Study IDs: 16-448; P50CA127003 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
This research study is looking at people with cancer of the pancreas to find clinical factors that can explain the presence of genetic mutations

DETAILED DESCRIPTION:
This research is being done to identify which pancreatic cancer patients should undergo genetic evaluation. A patient's personal and family history of cancer is the information typically used to make this decision, but there are currently no accurate, evidence-based guidelines that exist to help doctors use this information to make a decision.

The investigators hope that by testing all new pancreatic cancer patients, they can determine which clinical factors predict for genetic mutations in order to create a risk assessment tool.

The investigators want to determine which patients with pancreatic cancer will benefit from genetic testing. To do so, the investigators will offer all patients with pancreatic cancer in the Dana-Farber Gastrointestinal Oncology clinic referral for genetic evaluation. At the Cancer Genetics and Prevention clinic appointment, the provider will review the patient's personal and familial history of cancer and offer genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic ductal adenocarcinoma
* Signed initial informed consent
* Participant agrees to genetic counseling

Exclusion Criteria:

* Prospective participant unable to sign informed consent based on referring physician recommendation.
* Patient has neuroendocrine pancreatic tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient seen at Dana Farber Cancer Institute with a diagnosis of pancreatic ductal adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
We will measure clinical factors (e.g. # of PDAC patients with a personal history of x,y,z; # of PDAC patients with a family history of x,y,z; # PDAC patients with a germline mutation in x,y,z) so as to develop a risk assessment tool | Up to 5 years

SECONDARY OUTCOMES:
Evaluate Patient Experience With Genetic Testing | up to 5 years
Summarize patient satisfaction with Genetic counseling | up to 5 years
Number of patients who disclose genetic testing results to relatives | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Yurgelun, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No